CLINICAL TRIAL: NCT05499858
Title: Evaluating Effectiveness of Spices and Herbs to Increase Vegetable Intake Among Military
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: University of Maryland, Baltimore (Other); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); Pennington Biomedical Research Center (Other); McCormick Science Institute (Industry)
Responsible Party: Principal Investigator, Jonathan Scott, Assistant Professor, Uniformed Services University of the Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: USUHS- 2022-105
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Dietary Intake
Keywords: Military; Vegetable intake; Food photography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vegetables (Other): Vegetables will be provided to volunteers as part of a heat and serve meal kit.
  Interventions: Other: Spiced; Other: Plain

INTERVENTIONS:
Other: Spiced — Vegetables provided to volunteers will be spiced.
Other: Plain — Vegetables provided to volunteers will be plain.

SUMMARY:
"The goal of this study is to evaluate whether the addition of spices and herbs to the vegetables served to military personnel on a large military base can increase vegetable intake as compared to typical vegetable offerings without spices and herbs.

A two-phase intervention will be conducted on base at Naval Station Activity Bethesda (NSAB) to evaluate whether the addition of spices and herbs to vegetable dishes can increase vegetable intake amongst military service members.

Phase I will involve extensive engagement with key stakeholders involved in current vegetable consumption at NSAB, including military service members, staff dietitians, the health promotion specialist on base, barracks managers, military culinary specialist, unit leaders, morale welfare and recreations/single sailor program leaders, base senior enlisted leaders, and the base commander. Questionnaires will be administered evaluating current barriers to vegetable intake at NSAB, familiarity with and liking of a variety of spices and herbs, and sensory testing of several vegetables with and without spices and herbs. The recipes in the vegetable sensory testing comparisons will be identical other than spices and herbs content.

Phase II will involve will focus upon the direct measurement of vegetable intake (primary outcome) and vegetable linking (secondary outcome) among active-duty service members with spices and herbs and without spices and herbs. The vegetables will be provided as part of an entire meal on a "grab and go" plate. The other foods in the meal (proteins, starches, etc.) accompanying the vegetables will be kept consistently paired to vegetable recipes to minimize confounding. Vegetable intake will be assessed via cell phone pictures and liking will be assessed by a single 5-point Likert scale question."

ELIGIBILITY:
Inclusion Criteria:

* Junior Service Member (E1-E4 or O1-O3)
* Read and write English

Exclusion Criteria:

* Anyone under 18 years of age
* Anyone not in the U.S. military

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-11-06 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Vegetable consumption | Volunteers will be provided with a series of heat and serve meal kits over approximately 2 month time period.
  Volunteers will provided with a heat and serve meal kit. Using the food photography mobile application (SmartIntake), volunteers will take a single photo of the meal kit after they have consumed a self-determined desired amount of food. The digital photo will be sent to Pennington Biomedical Research Center (PBRC) for analysis via the SmartIntake app. The team at PBRC will download the image and use a validated algorithm to estimate, in cups, the remaining vegetable component from the meal kit.
Phase I - Primary Outcome: United States Military - Menu Item Survey | Volunteers will be provided with a series of 8 recipes to evaluate over the course of a single taste testing session through study completion, an average of 1 year.
  Overall liking of menu item, specific ratings of the appearance, aroma, flavor, texture, and overall appeal of the menu item, and qualitative feedback on general impressions of the menu item

CONTACTS AND LOCATIONS:
Overall Officials: Chris D'Adamo, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Naval Support Activity Bethesda, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No Personal Identifiable Information (PII) will be collected. All results will be deidentified and analyzed in aggregate.

REFERENCES:
- [Background] D'Adamo CR, McArdle PF, Balick L, Peisach E, Ferguson T, Diehl A, Bustad K, Bowden B, Pierce BA, Berman BM. Spice MyPlate: Nutrition Education Focusing Upon Spices and Herbs Improved Diet Quality and Attitudes Among Urban High School Students. Am J Health Promot. 2016 May;30(5):346-56. doi: 10.1177/0890117116646333. PMID 27404643
- [Background] Pierce B, Bowden B, McCullagh M, Diehl A, Chissell Z, Rodriguez R, Berman BM, D Adamo CR. A Summer Health Program for African-American High School Students in Baltimore, Maryland: Community Partnership for Integrative Health. Explore (NY). 2017 May-Jun;13(3):186-197. doi: 10.1016/j.explore.2017.02.002. Epub 2017 Feb 24. PMID 28373062
- [Background] D'Adamo CR, Parker EA, McArdle PF, Trilling A, Bowden B, Bahr-Robertson MK, Keller KL, Berman BM. The addition of spices and herbs to vegetables in the National School Lunch Program increased vegetable intake at an urban, economically-underserved, and predominantly African-American high school. Food Qual Prefer. 2021 Mar;88:104076. doi: 10.1016/j.foodqual.2020.104076. Epub 2020 Sep 1. PMID 32999533